CLINICAL TRIAL: NCT04378023
Title: Liver Transplant Combined With Neoadjuvant Chemo-radiotherapy in the Treatment of Unresectable Hilar Cholangiocarcinoma. A Prospective Multicenter Study.
Status: Recruiting | Type: Observational
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Cristina Dopazo Taboada, Consultant Surgeon, Hospital Vall d'Hebron
Other Study IDs: hCCA-LT
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Unresectable Cholangiocarcinoma
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients with unresectable hilar cholangiocarcinoma (hCCA) ≤3cm in radial diameter, without evidence of lymph node or distant metastases
  Interventions: Drug: Neoadjuvant Chemo-radiotherapy; Procedure: Liver Transplantation

INTERVENTIONS:
Drug: Neoadjuvant Chemo-radiotherapy — Patients will receive neoadjuvant radiotherapy (External - 50-54 grays) following by concomitant oral capecitabine (825mg/m2 bid).Thereafter, gemcitabine iv (1000mg/m2) plus cisplatin iv (25mg/m2) will be administered the day 1 and 8 every 21 days until transplant.
Procedure: Liver Transplantation — If no spread disease is discovered after neoadjuvant treatment, the patient will be listed for liver transplantation.

SUMMARY:
A prospective multicentre study which includes patients ≤ 70 years-old diagnosed of unresectable hilar cholangiocarcinoma (hCCA) ≤3cm in radial diameter, without evidence of lymph node or distant metastases. Liver transplantation preceded by neoadjuvant radio-chemotherapy will be performed in this selected group.

The primary endpoint will be overall survival at 1, 3, and 5 years post-transplant. The secondary endpoints will be: 1) recurrence free survival at 1, 3 and 5 years post-transplant; 2) intention-to-treat survival of overall patients included in the study at 1,3 and 5 year; 3) the rate of patients included in the study who are finally transplanted.

DETAILED DESCRIPTION:
A prospective multicentre pilot study which includes patients ≤ 70 years-old diagnosed of unresectable hilar cholangiocarcinoma (hCCA) ≤3cm in radial diameter, without evidence of lymph node or distant metastases.

The number of subjects necessary is 34 patients to achieve a power of 82% with a significance level of 0.05 to detect a 40% difference between the estimated 50% survival of those patients who are transplanted and 10% of those patients with hCCA unresectable who are not transplanted. This corresponds to a hazard ratio of 3.3219. Estimated loss to follow-up of 10% of patients.

RADIOLOGICAL EVALUATION

It will be considered unresectable those lesions Bismuth IV with the following criteria (Jarnagin WR, et al. Ann Surg 2001; 234:507; Memorial Sloan Kettering Cancer Center Hilar Cholangiocarcinoma Classification):

* Bilateral extension to second order biliary
* Unilateral extension to second-order biliary radicals AND contralateral portal vein involvement OR contralateral hepatic lobar atrophy
* Main or bilateral portal vein involvement
* Insufficient future liver remnant even after portal embolization

It will be performed the tumoral marker (CA 19.9), multiphase chest-abdomen CT scan, magnetic resonance cholangiopancreatography (MRCP) as well as positon emission tomography (PET)-scan if there is doubts of distant disease and upper endoscopic ultrasound (EUS) in order to rule out any obvious lymph node metastases. A biliary drainage will be placed by percutaneous transhepatic biliary drainage (PTBD) or endoscopic biliary drainage (EBD).

NEOADJUVANT TREATMENT

Patients will receive neoadjuvant radiotherapy (External - 50-54 grays) following by concomitant oral capecitabine (1,330mg/m2).Thereafter, gemcitabine iv (1000mg/m2) plus cisplatin iv will be administered the day 1 and 8 every 21 days until transplant.

A staging laparotomy/laparoscopy is recommended before including the patient in waiting list for transplant to confirm the abscence of extra-hepatic disease, especially peritoneal seeding and lymph nodes involvement.

A score exception will be allowed to optimized the treatment received and to be transplanted during the first 6 months.

LIVER TRANSPLANT AND FOLLOW UP

Regarding liver transplant technique, hepatic artery should be avoided for arterial reconstruction using the splenic artery or an iliac conduit.

Biomarker analyses in the explant specimen will be performed.

The patient will be monitored post-operatively at the clinical, biological and morphological levels every 3 months during the first 2 years and every 6 months thereafter in order to detect any recurrence and in the context of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written consent form
* Age ≤ 70 years-old
* ECOG 0 or 1
* Unresectable hCCA ≤3cm in radial diameter

Exclusion Criteria:

* Those patients who have received chemotherapy or radiotherapy previously out of protocol
* Liver, extrahepatic or lymph node metastases
* Previous intent of surgical resection or percutaneous biopsy
* Previous or concurrent cancer that is different in primary site or histology from adenocarcinoma, except cervical carcinoma in situ, localized prostate cancer, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, T1). Any cancer curatively treated 5 years prior to entry is permitted.
* Infection no controlled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients with unresectable malignant appearing hilar stricture and at least one of the following:
  * Malignant cytology or histology
  * CA 19.9>130U/mL without cholangits or/and jaundice
  * Mass on cross-sectional imaging
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 1, 3, and 5 years post-transplant | 5 years

SECONDARY OUTCOMES:
Recurrence free survival at 1, 3 and 5 years post-transplant | 5 years
Intention-to-treat survival of overall patients included in the study at 1,3 and 5 year | 5 years
The rate of patients included in the study who are finally transplanted. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Dopazo, Principal Investigator — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA, BARCELONA; Ramón Charco-Torra, Principal Investigator — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA, BARCELONA; Sonia Pascual-Bartolomé, Study Chair — HOSPITAL GENERAL UNIVERSITARIO, ALICANTE; Carmelo Loinaz-Segurola, Study Chair — HOSPITAL UNIVERSITARIO 12 DE OCTUBRE, MADRID; José María Álamo-Martinez, Study Chair — HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO, SEVILLA; José Luis Lucena de la Poza, Study Chair — HOSPITAL UNIVERSITARIO PUERTA DE HIERRO, MAJADAHONDA; Arturo Colon-Rodríguez, Study Chair — HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARANON, MADRID; Diego López-Segarra, Study Chair — COMPLEJO HOSPITALARIO UNIVERSITARIO, BADAJOZ; Yilliam Fundora-Suárez, Study Chair — Hospital Clinic of Barcelona; Andrea Bosca-Robledo, Study Chair — Hospital Universitario La Fe; Juan Andrés Echeverri-Cifuentes, Study Chair — HOSPITAL UNIVERSITARIO MARQUES DE VALDECILLA, SANTANDER; Marina Vila-Tura, Study Chair — HOSPITAL UNIVERSITARIO DE BELLVITGE, BARCELONA; Xavier Merino-Casabiel, Study Chair — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA, BARCELONA; David Leiva-Pedraza, Study Chair — HOSPITAL UNIVERSITARIO DE BELLVITGE, BARCELONA; María Teresa Salcedo-Allende, Study Chair — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA, BARCELONA; José Antonio Gracia Solanas, Study Chair — HOSPITAL CLÍNICO UNIVERSITARIO LOZANO BLESA, ZARAGOZA; Manuel Angel Barrera-Gómez, Study Chair — HOSPITAL UNIVERSITARIO NUESTRA SEÑORA DE LA CANDELARIA, TENERIFE; Ricardo Robles-Campos, Study Chair — Hospital Universitario Virgen de la Arrixaca; Laura Lladó-Garrida, Study Director — HOSPITAL UNIVERSITARIO DE BELLVITGE, BARCELONA; María Teresa Macarulla-Mercadé, Study Director — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA DE BARCELONA; Begoña Navalpotro-Yagüe, Study Director — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA DE BARCELONA; Florian Castet, Study Chair — HOSPITAL UNIVERSITARIO VALL D´HEBRON, UNIVERSIDAD AUTONOMA DE BARCELONA; Julio Santoyo, Study Chair — HOSPITAL REGIONAL UNIVERSITARIO DE MALAGA; Manuel Durán Martínez, Study Chair — HOSPITAL UNIVERSITARIO REINA SOFIA DE CÓRDOBA; Natalia Zambudio, Study Chair — Hospital Virgen de las Nieves (Granada)
Locations (1):
- Department of HPB Surgery and Transplants, Hospital Vall d´Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jarnagin WR, Fong Y, DeMatteo RP, Gonen M, Burke EC, Bodniewicz BS J, Youssef BA M, Klimstra D, Blumgart LH. Staging, resectability, and outcome in 225 patients with hilar cholangiocarcinoma. Ann Surg. 2001 Oct;234(4):507-17; discussion 517-9. doi: 10.1097/00000658-200110000-00010. PMID 11573044
- [Result] Heimbach JK, Gores GJ, Haddock MG, Alberts SR, Nyberg SL, Ishitani MB, Rosen CB. Liver transplantation for unresectable perihilar cholangiocarcinoma. Semin Liver Dis. 2004 May;24(2):201-7. doi: 10.1055/s-2004-828896. PMID 15192792
- [Result] Rea DJ, Heimbach JK, Rosen CB, Haddock MG, Alberts SR, Kremers WK, Gores GJ, Nagorney DM. Liver transplantation with neoadjuvant chemoradiation is more effective than resection for hilar cholangiocarcinoma. Ann Surg. 2005 Sep;242(3):451-8; discussion 458-61. doi: 10.1097/01.sla.0000179678.13285.fa. PMID 16135931
- [Result] Darwish Murad S, Kim WR, Harnois DM, Douglas DD, Burton J, Kulik LM, Botha JF, Mezrich JD, Chapman WC, Schwartz JJ, Hong JC, Emond JC, Jeon H, Rosen CB, Gores GJ, Heimbach JK. Efficacy of neoadjuvant chemoradiation, followed by liver transplantation, for perihilar cholangiocarcinoma at 12 US centers. Gastroenterology. 2012 Jul;143(1):88-98.e3; quiz e14. doi: 10.1053/j.gastro.2012.04.008. Epub 2012 Apr 12. PMID 22504095
- [Result] Ethun CG, Lopez-Aguiar AG, Anderson DJ, Adams AB, Fields RC, Doyle MB, Chapman WC, Krasnick BA, Weber SM, Mezrich JD, Salem A, Pawlik TM, Poultsides G, Tran TB, Idrees K, Isom CA, Martin RCG, Scoggins CR, Shen P, Mogal HD, Schmidt C, Beal E, Hatzaras I, Shenoy R, Cardona K, Maithel SK. Transplantation Versus Resection for Hilar Cholangiocarcinoma: An Argument for Shifting Treatment Paradigms for Resectable Disease. Ann Surg. 2018 May;267(5):797-805. doi: 10.1097/SLA.0000000000002574. PMID 29064885